CLINICAL TRIAL: NCT04786860
Title: The Success Rate of Cardiopulmonary Resuscitation in Patients Experiencing In-hospital Cardiac Arrest at Sanglah General Hospital
Brief Title: The Success Rate of Cardiopulmonary Resuscitation in Patients Experiencing In-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, MD, Principal Investigator, Udayana University
Other Study IDs: UNUD-CTR-FK210321-001
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrest, Sudden; Cardiopulmonary Arrest; Cardiopulmonary Failure; In-hospital Cardiac Arrest
Keywords: in-hospital, cardiac arrest, resuscitation, success rate
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CPR — Cardiopulmonary resuscitation performed on patients with in-hospital cardiac arrest

SUMMARY:
Cardiac arrest causes the heart to stop functioning to maintain circulation that provides oxygen to the brain. The global incidence of cardiac arrest is 50 to 60 per 100,000 people per year. The incidence of cardiac arrest in Indonesia in 2016 was 350,000 cases, in which 12% were successfully resuscitated, compared to the global success rate of 24.8%.

Cardiac arrest events urgently require CPR action that is useful to save lives in an emergency. The application of Code Blue aims to reduce the mortality rate and increase the rate of return of spontaneous circulation. The Code Blue team itself includes a set of teams who are trained in the handling of cardiorespiratory arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with in-hospital cardiac arrest that were treated at Sanglah General Hospital

Exclusion Criteria:

* Patients who upon admission to the hospital already showing cardiac arrest rhythm
* Patients who were DOA (death-on-arrival)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Survivors | 6-hours after CPR is stopped
  The number of patients who were successfully converted to ROSC (return of spontaneous circulation)

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Prof. Ngoerah General Hospital, Denpasar, Bali
  - Sanglah General Hospital, Denpasar, Bali

IPD SHARING:
Plan to Share IPD: Undecided